CLINICAL TRIAL: NCT02049658
Title: The Sensitivity and Specificity of Sniff Dog as a Tool in Diagnosing the Suspected Tumor Patients
Status: Recruiting | Type: Observational
Sponsor: Chang-Qing Gao (Other)
Responsible Party: Sponsor-Investigator, Chang-Qing Gao, MD PhD, Central South University
Organization: Central South University (Other)
Other Study IDs: Xiang-Ya 0003; XY 0003
Record Dates: First submitted 2014-01-26; First posted 2014-01-30 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Neoplasia
Keywords: tumor; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy volunteers: Healthy volunteers measured by currently used healthy screening procedures
- Suspected breast cancer subjects: Suspected breast cancer subjects without pathological examination yet but will have it soon
- Suspected lung cancer subjects: Suspected lung cancer subjects without pathological examination yet but will have it soon
- Suspected neurological tumor subjects: Suspected neurological tumor subjects without pathological examination yet but will have it soon
- Suspected patients with gynecological tumor: Suspected subjects with gynecological tumors without pathological examination yet but will have it soon

SUMMARY:
Previous studies have demonstrated that sniff dogs can identify cancer patients from healthy subjects through sniffing exhaled breath air or blood or serum or urine or feces. It is hypothesized that sniff dogs may be used as a tool in identifying cancer patients in the high risk population or suspected patients. Trained dogs will sniff serum from participants who are suspected to suffer from tumor by their physicians and not yet but will be diagnosed by pathological examination.The results will be compared with the outcome of the pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who have been examined by the currently used procedures and find to be without tumors.
* Patients in the breast surgery, thoracic surgery, gynecological and neurosurgery departments with lesions with characteristics of tumors

Exclusion Criteria:

* Patients who have had pathological results

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Healthy volunteers who have been examined by the currently used procedures and find to be without tumors.
  * Patients in the breast surgery, thoracic surgery, gynecological and neurosurgery departments with lesions with characteristics of tumors
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of the sniff dogs as a tool in diagnosing tumors | 12 months
  The results that obtained from the dogs will be compared with these of the pathological examinations. Sensitivity = the No. of patients identified by the dogs as cancers / the No. of patients suffering from cancer confirmed by pathological examination. Specificity = No. of subjects signaled by the dog as non-cancers / No. of subjects confirmed by pathological examination as non-cancer subjects.

SECONDARY OUTCOMES:
behavior patterns of the sniff dogs to different diseases | 12 months
  The behavior (lying before the tank for positive, neglecting the tanks) of the dog will be recorded and compared with the results of the pathological examination.

OTHER OUTCOMES:
the substances used for identifying tumors by the sniff dogs | 12 months
  GCMS etc will be used to compare the volatile compounds between the sera from cancers patients and the from non-cancer subjects, the suspected VOCs will be tested by the dog for conformation.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Qing Gao, MD PhD, Principal Investigator — Central South University
Locations (1):
- Center for Scientific Research with Animal Models, CSU, Changsha, Hunan, China